CLINICAL TRIAL: NCT06553287
Title: A Phase Ib, Randomized, Double-Blind, Vehicle-Controlled, Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LNK01004 Ointment in Adults Patients With Mild to Moderate Atopic Dermatitis.
Brief Title: Safety, Tolerability and Pharmacokinetics of LNK01004 Ointment in Adults With Atopic Dermatitis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lynk Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LK004102
Record Dates: First submitted 2024-08-10; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LNK01004 ointment 0.3% (Experimental): Participants will receive LNK01004 ointment 0.3% twice daily
  Interventions: Drug: LNK01004 ointment 0.3%
- LNK01004 ointment 1.0% (Experimental): Participants will receive LNK01004 ointment 1.0% twice daily
  Interventions: Drug: LNK01004 ointment 1.0%
- LNK01004 ointment 1.5% (Experimental): Participants will receive LNK01004 ointment 1.5% twice daily
  Interventions: Drug: LNK01004 ointment 1.5%
- Vehicle (Experimental): Participants will receive vehicle BID
  Interventions: Drug: Vehicle BID

INTERVENTIONS:
Drug: LNK01004 ointment 0.3% — LNK01004 ointment 0.3% for topical application
  Arms: LNK01004 ointment 0.3%
Drug: LNK01004 ointment 1.0% — LNK01004 ointment 1.0% for topical application
  Arms: LNK01004 ointment 1.0%
Drug: LNK01004 ointment 1.5% — LNK01004 ointment 1.5% for topical application
  Arms: LNK01004 ointment 1.5%
Drug: Vehicle BID — Inactive vehicle matched to LNK01004 ointment for topical application.
  Arms: Vehicle

SUMMARY:
The purpose of the study is to evaluate the Safety, Tolerability, and Pharmacokinetics of LNK01004 ointment (0.3%, 1.0%, and 1.5%) vs vehicle twice daily (BID) in Adults Patients with Atopic Dermatitis.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, vehicle-controlled, dose-escalation study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LNK01004 ointment twice daily (BID) in participants with Mild to Moderate atopic dermatitis as compared with vehicle cream BID.

ELIGIBILITY:
Inclusion Criteria:

* Participants were diagnosed with atopic dermatitis (AD) for at least 6 months.
* Participants with an Investigator's Global Assessment (IGA) score of 2 to 3 at screening and baseline.
* Participants with body surface area (BSA) of AD involvement, excluding the scalp, face, and intertriginous areas, of 3% to 20% at screening and baseline.
* BMI of 18.0-30.0 kg/m2, with body weight ≥ 50 kg for man and ≥ 40 kg for woman.
* Be willing to comply with the study lifestyle restraints, e.g., no washing of the administered area within 6 hours of study drug administration, no sweaty exercise.

Exclusion Criteria:

* Participants with a physical condition which, in the Investigator´s opinion, might interfere with the assessment of atopic dermatitis or expose the patient to an unacceptable risk by study participation.
* Participants with current evidence of any acute skin infection with a history of recurrent or chronic severe skin infection.
* Participants with known allergies to components or excipients of the test drug.
* Participants who are pregnant, nursing, or planning a pregnancy during the study period.
* Systemic immunosuppressive or immunomodulating drugs (eg, oral or injectable corticosteroids, mycophenolate mofetil, PDE4 inhibitor) used for atopic dermatitis within 4 weeks or 5 half-lives of baseline (whichever is longer).
* Participants with the following hematologic abnormities at screening:
* Leukocytes < 3.0 × 10^9/L.
* Neutrophils < lower limit of normal.
* Hemoglobin < 10 g/dL.
* Lymphocytes < 0.8 × 10^9/L
* Platelets < 100 × 10^9/L.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 1.5 × upper limit of normal.
* TBiL ≥ 1.5 × ULN, or ULN < TBiL < 1.5 × ULN but judged by the investigator to be abnormal clinically significant;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events (TEAE) | Baseline up to week 4
  Number of participants with at least one TEAE.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) for LNK01004 in plasma | Day1 and Day 7
  Cmax is defined as the maximum observed plasma concentration for LNK01004
Area under plasma concentration versus time curve, time zero to infinity | Day 1 and Day7
  The area under the plasma concentration-time curve is a method of measurement of the total exposure of a drug in plasma
Mean Percentage Change From Baseline in Eczema Area and Severity Index (EASI) Score | Baseline and Weeks 1, 2, and 4
  The EASI is an instrument to measure the severity and extent of AD. The body is first divided into 4 areas: head (10% of skin), arms (20%), trunk (30%), and legs (40%). Then, the area affected is scored from 0 (0% involvement) to 6 (90-100% involvement), and severity is scored from 0 ('none') to 3 ('severe'). The EASI combines the area affected and severity ratings to get a final composite score ranging from 0 (no disease) to 72 (maximal disease). Note that palms and soles were treated as appropriate but were not counted towards any measurements of EASI.
Number of Participants Achieving a 75% Decrease From Baseline in EASI Score (EASI-75) | Baseline and Weeks 1, 2, and 4
  The number of participants with a decrease of at least 75% from the baseline EASI total score is presented. The EASI is an instrument to measure the severity and extent of AD. The body is first divided into 4 areas: head (10% of skin), arms (20%), trunk (30%), and legs (40%). Then, the area affected is scored from 0 (0% involvement) to 6 (90-100% involvement), and severity is scored from 0 ('none') to 3 ('severe'). The EASI combines the area affected and severity ratings to get a final composite score ranging from 0 (no disease) to 72 (maximal disease), with positive results indicating an increase from baseline in EASI total score (i.e., increased symptoms) and negative results indicating a decrease from baseline score (i.e., decreased symptoms). Note that palms and soles were treated as appropriate but were not counted towards any measurements of EASI.
Number of Participants Achieving ≥4-Point Improvement in WI-NRS Pruritus Score | Baseline and Weeks 1, 2, and 4
  The number of participants achieving a ≥4-point improvement from Baseline in WI-NRS score is presented. The WI-NRS is a simple, single item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the subject experienced in the previous 24 hours. Higher scores indicate greater symptom severity.
Percentage of Participants Achieving an Investigator's Global Assessment (IGA) Score of 0 to 1 Who Have an Improvement of ≥ 2 Points From Baseline | Baseline and Weeks 1, 2, and 4
  IGA is an assessment scale used to determine severity of atopic dermatitis (AD) and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear). An IGA responder was defined as a participant achieving an IGA score of 0 to 1 and an IGA score improvement at least 2 from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Qianjin Lu, Principal Investigator — Hospital for skin diseases, Institute of Dermatology, Chinese Academy of Medical Sciences.
Locations (1):
- Hospital for skin diseases, Institute of Dermatology, Chinese Academy of Medical Sciences., Nanjing, China